CLINICAL TRIAL: NCT01988532
Title: Impact of Pain on Functional Impairment and Quality of Life in Adults With Hemophilia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-4073; U1111-1138-3464 (Other: WHO)
Record Dates: First submitted 2013-10-17; First posted 2013-11-20 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia A With Inhibitors; Haemophilia B; Haemophilia B With Inhibitors
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult PWH
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will only fill out a questionnaire

SUMMARY:
This study is conducted in the United States of America (USA). The aim of the study is to assess the impact of pain on functional impairment and quality of life in adult persons with hemophilia (PWH) with and without inhibitors with joint bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Adult males able to provide consent and complete a survey in English
* Congenital hemophilia A or B with or without inhibitors with any history of joint bleeding or joint pain
* Presentation at the treatment center for a comprehensive annual visit where joint range of motion will be obtained
* Informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol)

Exclusion Criteria:

* Previous participation in this study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult PWH in the United States of America (USA) willing to consent to participation who have any history of joint bleeding or joint pain presenting for a comprehensive care visit during which joint range of motion will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute (bleed-related) pain (percentage) | At the first visit (only one study visit)
Prevalence of chronic (arthritic) pain (percentage) | At the first visit (only one study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- [Result] Wang M., Baumann K., Akins S., Funk S., Hernandez G., Kempton C., Buckner T., Cooper D. Pain, Functional Impairment, and Quality of Life (P-FIQ): Reliability of Patient-Reported Outcome (PRO) Instruments Assessing Pain and Function in US Adult People With Hemophilia (PWH). 14th WFH International Musculoskeletal Congress 2015; : Abstract number: P-224 Country: Northern Ireland City: Belfast
- [Result] Baumann K., Akins S., Funk S., Hernandez G., Kempton C., Wang M., Buckner T., Cooper D. Functional Impairment, Pain, and Pain Management in Adult People with Haemophilia (PWH): Initial Lessons from the Pain Functional Impairment and Quality of Life (P-FIQ) Study. 14th WFH International Musculoskeletal Congress 2015; : Abstract number: MP-209 Country: Northen Ireland City: Belfast
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com